CLINICAL TRIAL: NCT06613360
Title: A Phase 1b, Open-label, Pilot Study of CLN-978 for the Treatment of Moderate to Severe Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of CLN-978, a Subcutaneously Administered CD19-directed T Cell Engager, in Subjects With Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cullinan Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLN-978-SL-101
Record Dates: First submitted 2024-09-20; First posted 2024-09-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: SLE; SLE (Systemic Lupus)
Keywords: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A Dose Escalation (Experimental): Patients with SLE treated with CLN-978 in dose escalation cohorts
  Interventions: Drug: CLN-978
- Part B Further Dose Evaluation (Experimental): Further evaluation of CLN-978 treatment of patients with SLE
  Interventions: Drug: CLN-978

INTERVENTIONS:
Drug: CLN-978 — Specified dose on specified days

SUMMARY:
Phase 1b, open-label study of CLN-978 administered subcutaneously in patients with Moderate to Severe Systemic Lupus Erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE at least 24 weeks prior to Screening and meet 2019 EULAR / ACR Classification Criteria at screening.
* Presence of one or more of the following autoantibodies documented during screening or in the previous 12 months before screening: positive anti-nuclear antibody (ANA) test (≥1:80); anti dsDNA above the upper limit of normal (ULN); anti-Sm above the ULN.
* Active SLE disease, as demonstrated by a SLEDAI total score ≥6 at screening.
* Inadequate response to at least 2 of the following treatments: oral corticosteroid, antimalarials, conventional immunosuppressants, or biologics. At least one of the failed treatments should be an immunosuppressive or biologic standard-of care agent.
* If on corticosteroid and/or antimalarial, the dose must be stable prior to day 1.
* Laboratory parameters including the following:

  * Absolute lymphocyte count (ALC) ≥0.5 x 109/L
  * Peripheral B cell count ≥25 cells/µL
  * Absolute neutrophil count (ANC) ≥1.0 x 109/L
  * Hemoglobin ≥8 g/dL
  * Platelet count ≥75 x 109/L.
  * Estimated glomerular filtration rate (eGFR) (based on CKD-EPI formula) ≥30 mL/min/1.73m2
  * Total bilirubin ≤1.5 × ULN, except patients with confirmed Gilbert's Syndrome
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN
* Part B only: For patients who were treated in Part A and did not experience dose-limiting toxicity (DLT) or discontinue CLN-978 treatment due to AEs are eligible for retreatment at a higher dose or longer schedule in Part B if they otherwise meet eligibility criteria and at least 90 days have passed since the last dose of CLN-978.

Exclusion Criteria:

* Active inflammatory disease other than SLE. Thyroiditis or secondary Sjogren's syndrome is allowed.
* Considered at high risk for thrombosis.
* Rapidly progressive glomerulonephritis, and/or urine protein/creatinine >3 mg/mg (339 mg/mmol).
* Active severe neuropsychiatric/CNS manifestations of SLE.
* Evidence of hepatitis B, hepatitis C (HCV) infection, human immunodeficiency virus (HIV), Epstein-Barr virus (EBV), or cytomegalovirus (CMV) infection.
* History of splenectomy.
* Prior treatment with the following:

  * Cellular or gene therapy product directed at any target.
  * Investigational therapy within 30 days or 5 drug-elimination half-lives (whichever is longer) prior to Day 1.
  * Any anti-CD19 or anti-CD20 therapy less than 3 months prior to Day 1.
  * Non-biologic DMARD within 14 days prior to Day 1.
  * Cyclophosphamide within 1 month or a biologic immunomodulating therapy during 2 months prior to Day 1.
* Live or attenuated vaccine within 28 days prior to screening or during screening.
* Active, clinically significant bacterial, viral, fungal, mycobacterial, parasitic, or other infection, including SARS-CoV-2 infection, within 14 days before Day 1.
* Active or latent tuberculosis (TB) evidenced by a positive or indeterminant Interferon Gamma Release Assay (IGRA), unless the patient has documented previous completion of TB treatment and no current clinical indication of TB.
* Any condition for which, in the opinion of the Investigator and/or Sponsor, would not be in the best interest of the patient to participate in the study or that could prevent, limit, or confound any protocol-defined assessment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 48 weeks
  Incidence and severity of adverse events (AEs)/adverse events of special interest (AESIs)/serious adverse events (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetics | 48 weeks
  Serum concentrations of CLN-978
Immunogenicity | 48 weeks
  Level of anti-drug antibodies
Pharmacodynamics-related biomarker | 48 weeks
  Levels of total B lymphocytes in the peripheral blood

OTHER OUTCOMES:
hybrid Systemic Lupus Erythematosus Disease Activity Index (hSLEDAI) | 48 weeks
  Change in hybrid Systemic Lupus Erythematosus Disease Activity Index (hSLEDAI) score on a scale of 0 to12 with a higher score meaning worse outcome
Physicians Global Assessment | 48 weeks
  Change in Physicians Global Assessment (PGA) score on a scale of 0 to 3 with a higher score indicating worse outcome

CONTACTS AND LOCATIONS:
Locations (14):
- United States (10):
  - Cullinan Investigative Site, Avondale, Arizona
  - Cullinan Investigative Site, Tucson, Arizona
  - Cullinan Investigative Site, Orlando, Florida
  - Cullinan Investigative Site, Iowa City, Iowa
  - Cullinan Investigative Site, New York, New York
  - Cullinan Investigative Site, Rochester, New York
  - Cullinan Investigative Site, Memphis, Tennessee
  - Cullinan Investigative Site, Plano, Texas
  - Cullinan Investigative Site, Webster, Texas
  - Cullinan Investigative Site, Salt Lake City, Utah
- Australia (2):
  - Cullinan Investigative Site, Parkville, Victoria
  - Cullinan Investigative Site, Victoria Park
- Arensia Research Clinic, Tbilisi, Georgia
- Arensia Research Clinic, Chisinau, Moldova